CLINICAL TRIAL: NCT05158686
Title: Use of Drug-Coated Balloon to Improve Recanalization of a Coronary Chronic Total Occlusion After Failed Angioplasty: The IMPROVED-RECTO Trial.
Brief Title: Use of Drug-Coated Balloon to Improve Recanalization of a Coronary Chronic Total Occlusion After Failed Angioplasty
Acronym: IMPROVED-RECTO
Status: Completed | Type: Observational
Sponsor: Ignacio J. Amat Santos (Other)
Responsible Party: Sponsor-Investigator, Ignacio J. Amat Santos, Coordinator of Interventional Cardiology Unit, Hospital Clínico Universitario de Valladolid
Organization: Hospital Clínico Universitario de Valladolid (Other)
Other Study IDs: ICICOR-IMPROVED-RECTO-2021
Record Dates: First submitted 2021-12-02; First posted 2021-12-15 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Chronic Total Occlusion
Keywords: Repeated procedure, Angioplasty, Paclitaxel, drug-coated balloon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Paclitaxel-coated balloon angioplasty: Patients with previous failed recanalization of a CTO treated with paclitaxel coated balloon immediately proximal to the CTO during the index procedure
  Interventions: Device: Paclitaxel-coated Balloon dilation angioplasty
- Non-coated balloon angioplasty: Patients with previous failed recanalization of a CTO treated with non-coated balloon immediately proximal to the CTO during the index procedure
  Interventions: Device: Non-coated Balloon dilation angioplasty

INTERVENTIONS:
Device: Paclitaxel-coated Balloon dilation angioplasty — Paclitaxel-coated ballon dilation angioplasty proximal to CTO lesion after failed percutaneous recanalization
  Groups: Paclitaxel-coated balloon angioplasty
Device: Non-coated Balloon dilation angioplasty — Non-coated ballon dilation angioplasty proximal to CTO lesion after failed percutaneous recanalization
  Groups: Non-coated balloon angioplasty

SUMMARY:
Observational retrospective registry to compare effectiveness of paclitaxel-coated vs. non coated balloon angioplasty proximal to a Chronic Total Occlussion (CTO) after failed revascularization. Primary objective is to determine success rate after repeated percutaneous coronary intervention of a CTO 3 to 6 months after paclitaxel-coated balloon angioplasty proximal to the persistent lesion.

ELIGIBILITY:
Inclusion Criteria:

* Failed recanalization of a CTO in patients with clinical indication for the percutaneous procedure.
* Patient willing to participate in the study providing signed informed consent.
* J-CTO Score ≥2.

Exclusion Criteria:

- Unfeasible recanalization of the CTO according to the interventional cardiologists of the center.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary angiography in which percutaneous coronary intervention results in failure during treatment of a CTO. Indication of the procedures will be clinically driven. Informed consent will be provided after the first failed attempt of CTO recanalization.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Success of repeated percutaneous coronary intervention of a CTO 3 to 6 months after balloon angioplasty proximal to the persistent lesion. | 6 months

SECONDARY OUTCOMES:
Mortality after second attempt of CTO recanalization | 6 months
Quality of life assessed by EQ5D questionnaire | 6 months
Procedural duration during second attempt | 6 months
Radiation during second attempt | 6 months
Contrast administration during second attempt | 6 months
Events at 1-year follow-up | 1 year
  All events including: Death, stroke, myocardial infarction (MI), target lesion revascularization (TLR), and contrast-induced nephropathy (CIN)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universitario de Valladolid, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No